CLINICAL TRIAL: NCT07132437
Title: Phase I Clinical Study of Systemic Pharmacokinetics and Safety of ZKY001 Eye Drops for Multiple Administration in Patients With Corneal Epithelial Defect After Corneal Endothelial Transplantation
Brief Title: Phase I Clinical Study of ZKY001 Eye Drops in the Treatment of Corneal Epithelial Defect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZKYK-ZKY001-DYD
Record Dates: First submitted 2021-09-17; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Corneal Diseases
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Intervention Model Description: A dose group of 0.004% was used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 0.004% ZKY001 eye drops (Experimental): Start taking the medicine from Day 1 and continue for 6 consecutive days.
  Interventions: Drug: ZKY001 EYE DROPS

INTERVENTIONS:
Drug: ZKY001 EYE DROPS — On the 1st postoperative day (Day1), ZKY001 eye drops were dropped into the experimental eyes (the operative eyes were taken as the experimental eyes). ZKY001 eye drops were given at 8:00 am ±1h from Day1 to Day5. 4 times a day, 1 drop each time, recommended interval of 4 to 6 hours.
  Day6 was administered at 8:00 am ±1h, and ZKY001 eye drops were dropped into the test eye (the surgical eye was taken as the test eye). Day6 was given only once, 1 drop each time.
  Other Names: Germinal peptide eye drops

SUMMARY:
One dose group of 0.004% was used.

DETAILED DESCRIPTION:
One dose group of 0.004% was used. The whole study includes two stages: pre-test and formal test.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-70 (including threshold);
2. Body mass index between 19-26kg/m2 (including critical value), male weight ≥50kg, female weight ≥45kg;
3. Patients who have undergone Descemet's stripping endothelial keratoplasty（DSEK）, Descemet's stripping automated endothelial keratoplasty（DSAEK） or Descemet membrane endothelial keratoplasty（DMEK） and need to remove corneal epithelium during surgery (the diameter of the removed epithelium area ≥8mm);
4. Lacrimal secretion test (Schirmer test I) ≥10mm/5min during screening;
5. Limbus structure was normal under slit-lamp during screening period;
6. Voluntarily sign informed consent.

Exclusion Criteria:

1. Smoking more than 5 cigarettes per day on average;
2. suspected or indeed alcohol dependence with an average intake of more than 2 units of alcohol per day for 3 months or positive alcohol test;
3. those who have a history of drug abuse or have a positive urine test;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Estimate pharmacokinetic parameters | Day 6
  Pharmacokinetic parameters（Area Under Curve from 0 to time t（AUC 0-t）） were estimated based on plasma concentration of ZKY001 after multiple dosing
Estimate pharmacokinetic parameters | Day 6
  Pharmacokinetic parameters（Area Under Curve from 0 to infinity（AUC 0-∞）） were estimated based on plasma concentration of ZKY001 after multiple dosing
Estimate pharmacokinetic parameters | Day 6
  Pharmacokinetic parameters（Area Under Curve at steady state（AUC ss）） were estimated based on plasma concentration of ZKY001 after multiple dosing
Estimate pharmacokinetic parameters | Day 6
  Pharmacokinetic parameters（Maximum Plasma Concentration（C max）） were estimated based on plasma concentration of ZKY001 after multiple dosing
Estimate pharmacokinetic parameters | Day 6
  Pharmacokinetic parameters（Minmum Plasma Concentration（C min）） were estimated based on plasma concentration of ZKY001 after multiple dosing
Estimate pharmacokinetic parameters | Day 6
  Pharmacokinetic parameters（Average Plasma Concentration（C av）） were estimated based on plasma concentration of ZKY001 after multiple dosing
Estimate pharmacokinetic parameters | Day 6
  Pharmacokinetic parameters（Degree of fluctuation（FD）） were estimated based on plasma concentration of ZKY001 after multiple dosing
Estimate pharmacokinetic parameters | Day 6
  Pharmacokinetic parameters（Maximum Time（T max）） were estimated based on plasma concentration of ZKY001 after multiple dosing
Estimate pharmacokinetic parameters | Day 6
  Pharmacokinetic parameters（half time（T 1/2）） were estimated based on plasma concentration of ZKY001 after multiple dosing
Estimate pharmacokinetic parameters | Day 6
  Pharmacokinetic parameters（apparent volume of distribution（Vd）） were estimated based on plasma concentration of ZKY001 after multiple dosing
Estimate pharmacokinetic parameters | Day 6
  Pharmacokinetic parameters（elimination rate constant（Kel）） were estimated based on plasma concentration of ZKY001 after multiple dosing
Estimate pharmacokinetic parameters | Day 6
  Pharmacokinetic parameters（Mean Residence Time（MRT）） were estimated based on plasma concentration of ZKY001 after multiple dosing
Estimate pharmacokinetic parameters | Day 6
  Pharmacokinetic parameters（Clearance（CL）） were estimated based on plasma concentration of ZKY001 after multiple dosing
Estimate pharmacokinetic parameters | Day 6
  Pharmacokinetic parameters（Clearance/Bioavailability（CL/F）） were estimated based on plasma concentration of ZKY001 after multiple dosing

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqiang Pan, Study Director — Beijing Tongren Hospital
Locations (1):
- Zhiqiang Pan, Beijing, China